CLINICAL TRIAL: NCT05755672
Title: On-treatment Biomarkers in Metastatic Colorectal Cancer for Life: The On-CALL Study
Brief Title: On-treatment Biomarkers in Metastatic Colorectal Cancer for Life
Acronym: On-CALL
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01242-01
Record Dates: First submitted 2023-02-17; First posted 2023-03-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Cancer; Chemotherapy Effect; Peritoneal Metastases; Liver Metastasis Colon Cancer; Lung Metastases
Keywords: Metastatic colorectal cancer; Chemotherapy; Targeted therapy; Tumor heterogeneity; Tumor evolution
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — * Tissue from the first histological specimen for diagnosis (usually a biopsy)
  * Blood sample during ongoing neoadjuvant and/or adjuvant chemotherapy
  * Tissue from the surgical resection specimen (primary tumour and resected metastases)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Synchronous mCRC patients: Patients diagnosed with synchronous metastatic colorectal cancer with planned treatment with curative intent at Skåne University Hospital (Malmö and Lund), who have accepted the study invitation (agreeing to participation - informed consent)
  Interventions: Drug: Chemotherapy; Procedure: Resection of the primary tumor; Procedure: Resection of tumour metastases; Procedure: Blood sampling during chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Neo-adjuvant and adjuvant chemotherapy with curative intent, according to the current clinical practice guidelines
Procedure: Resection of the primary tumor — Surgical resection of the primary tumour, according to the current clinical practice guidelines
  Other Names: Surgical resection of the primary tumour
Procedure: Resection of tumour metastases — Surgical resection of tumour metastases, according to the current clinical practice guidelines
  Other Names: Surgical resection of tumour metastases
Procedure: Blood sampling during chemotherapy — Drawing of blood samples several times during patient visits for chemotherapy regimen
  Other Names: Drawing of blood samples during chemotherapy

SUMMARY:
By virtue of an increased strategic use of cytotoxic and biological agents, and more options for locoregional treatment, the survival of patients with metastatic colorectal cancer (mCRC) has improved considerably in the past decades. The personalized approach to systemic treatment is further aided by the use of complementary molecular biomarkers. However, the evolutionary dynamics of mCRC, a disease harnessed by multiple adaptive genetic alterations towards its final stages, poses a particular challenge to single-sample biomarker analyses and standardized linear treatment protocols. The aim of the On-treatment biomarkers in metastatic ColorectAL cancer for Life (On-CALL) study is to generate further knowledge on the evolutionary progression of mCRC during treatment, and to elucidate the mechanisms underlying the therapeutic failure still seen in a substantial number of patients.

The On-CALL study is a prospective, single-arm observational study. All patients diagnosed with synchronous mCRC treated with curative intent at Skåne University Hospital will be invited to participate. Clinical and histopathological data will be compiled at study entry. An individual tissue microarray block with samples from resected primary tumours and metastases representing the full extent of the tumour spread will be constructed for each patient. Blood samples will be drawn for biomarker analyses at multiple time points prior to, during and after systemic treatment. DNA sequencing of tumour tissue and circulating tumour DNA (ctDNA) will be performed to define the spatial clonal landscape in primary tumours and metastases, as well as over time.

DETAILED DESCRIPTION:
The aim of the On-treatment biomarkers in metastatic ColorectAL cancer for Life (On-CALL) study is to generate further knowledge on the evolutionary progression of mCRC during treatment with curative intent, and to elucidate the mechanisms underlying the therapeutic failure still seen in a substantial number of patients.

The specific objectives are:

* To comprehensively characterise the spatial intertumoural, intermetastatic and intrametastatic genetic heterogeneity
* To delineate differences in the prevalence and type of genetic heterogeneity, as well as tumour evolvability, according to metastatic site
* To examine the associations between spatial and temporal heterogeneity
* To examine ctDNA quantity and quality as an early biomarker for response to neoadjuvant treatment
* To examine ctDNA quantity and quality as an early biomarker for response to adjuvant treatment
* To evaluate the relationship between phylogenetic patterns, i.e. the tumour evolvability, and survival in relation to different treatment modalities
* To examine the heterogeneity of the tumour microenvironment in relation to the genetic heterogeneity and evolvability of the tumours
* To examine circulating immune cells and inflammatory biomarkers, and their relationship with the genetic and microenvironmental heterogeneity of the tumours
* To delineate parallel events at the transcriptomic and proteomic levels, with particular reference to their potential utility as clinically relevant surrogate biomarkers of genetic alterations underlying the evolvability of the tumours

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of synchronous metastatic colorectal cancer, planned cancer treatment with curative intent at the Skåne University Hospital

Exclusion Criteria:

* Not accepting the study inclusion terms (informed consent not obtained)
* Age below or above the age limit

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are treated at the Skåne University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Follow-up examination of tumour remission, progression or recurrence | 10 years
  Radiological/clinical examination of tumour remission, progression or recurrence, and correlation of this clinical information with the available oncogenetic data from histological samples from the primary tumour and metastases, and from data from blood samples (ctDNA analysis)
  * Oncogenetic data will come from genomic profiling of tissue samples. This will be carried out by targeted deep sequencing (TDS), using a comprehensive panel covering cancer-related genes, in combination with genome wide SNP array for detection of copy number aberrations.
  * Data from blood samples will be extracted through quantification of ctDNA and monitoring of the temporal clonal dynamics (circulating cell free DNA will be extracted from plasma samples from all time points).

SECONDARY OUTCOMES:
Quality of life changes | 10 years
  Patients will take quality-of-life surveys (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - version EORTC-QLQ-C30 and EORTC-QLQ-CR29) will assistance of medical professionals prior to and after neoadjuvant and/or adjuvant treatment.
  * These surveys are cancer-specific core questionnaires for use in relation to various cancers.
  * The questionnaire scales the items on a score of 1 (Not at all) to 4 (Very much), and 1 (Very poor) to 7 (Excellent).
  * Scoring result is 0 to 100; for functional and global quality of life scales, higher scores mean a better level of functioning, and for symptom-oriented scales, a higher score means worse/more severe symptoms.
  * Statistical analysis will be performed with the data from the questionnaires, and the evolution/changes of symptoms and subjective experiences of the patients will be quantified and correlated with the clinical findings.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Jirström, M.D. PhD., Study Director — Region Skåne; Jakob Eberhard, M.D. PhD., Study Chair — Region Skåne
Locations (2):
- Sweden (2):
  - Department of Oncology, Hematology and Radiophysics, Skane University Hospital, Lund, Skåne County
  - Department of Oncology, Hematology and Radiophysics, Skane University Hospital, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: Undecided